CLINICAL TRIAL: NCT05463523
Title: Based on Artificial Intelligence, Augmented Reality and New Optical Imaging Technology, the Research and Development of a Skin Diseases Intelligent Diagnosis and Treatment System: A Multi-centric Clinical Trial in China
Brief Title: A Multi-centric Clinical Trial in China for Skin Diseases Intelligent Diagnosis and Treatment System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: XiangyaH001
Record Dates: First submitted 2021-12-09; First posted 2022-07-19 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2021-12

CONDITIONS: Skin Diseases; Artificial Intelligence; Augmented Reality; Medical Imaging
Keywords: Augmented Reality; Skin Tumor; Surgery Plan and Navigation; Dignosis and Treatment
MeSH Terms: conditions — Skin Diseases; Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Digital camera: A Real-time Augmented Reality Device with Artificial Intelligence Integration, acquisition of patient skin lesion images as data
  Interventions: Device: A Real-time Augmented Reality Device with Artificial Intelligence Integration

INTERVENTIONS:
Device: A Real-time Augmented Reality Device with Artificial Intelligence Integration — Patients are diagnosed and treated with the assistance of artificial intelligence, augmented reality and new optical imaging technology, which is different from traditional model.

SUMMARY:
In response to clinical needs, infrared multi-spectral images are combined with traditional clinical images and other multi-modal data to build a more efficient intelligent auxiliary diagnosis system and intelligent equipment for skin health and diseases, including skin lesions automatically segmentation on skin diseases images, automatically design surgical margin and planning for skin tumor surgery.

DETAILED DESCRIPTION:
Database: Relying on the preliminary foundation, build the first standardized infrared multispectral image database of skin diseases, and further integrate other medical images and medical history texts to iterate into a large multimodal skin disease database.

Model: Design a deep learning network based on multi-scale and multi-level. The collaborative attention learning network realizes the collaborative representation of multi-modal data at the feature level, builds a multi-modal skin disease auxiliary diagnosis model, and realizes breakthroughs in algorithms. Develop the segmentation network of skin lesions and model for surgery planning, including surgical margin design and navigation of intraoperative sampling.

System: Propose an artificial intelligence system combined with the real-time augmented reality to assist dignosis and surgery for skin diseases.

Equipment: Based on the self-developed high-performance system, construct and assemble infrared multi-spectral skin disease auxiliary diagnosis equipment and multifunctional device for skin tumors surgery.

ELIGIBILITY:
Inclusion Criteria:

* Informed consented.
* With a diagnosis of skin disease made by at least 3 dermatologists.
* Without life-threatening risk to intervention.
* Requires surgical treatment (For devices).

Exclusion Criteria:

* Having difficulties to follow-up.
* Poor general condition.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population is diagnosed of skin disease made by at least 3 dermatologists. For population who needs to use the system and device, requires surgical treatment and willing to underwent a new modality. Exclusions include poor general condition and having difficulties to follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Doctors' Evaluation | Give an evaluation immediately after using the system and equipment.
  Compare the proposed system's perfomance with the doctors in the terms of the diganosis and lesion segmentation. After using the system and the device, doctors evaluated its performance on the Skin Lesion Boundary Description, Margin Design, Sampling Navigation, Projection Effect, Security, Time-consuming and Convenience. 0-10 points for each indicator is scored independently by 4 doctors.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No